CLINICAL TRIAL: NCT01357161
Title: A Randomized, Phase II Study Evaluating MK-1775 in Combination With Paclitaxel and Carboplatin Versus Paclitaxel and Carboplatin Alone in Adult Patients With Platinum Sensitive p53 Mutant Ovarian Cancer
Brief Title: A Study of Adavosertib (MK-1775) in Combination With Paclitaxel and Carboplatin Versus Paclitaxel and Carboplatin Alone for Participants With Platinum-Sensitive Ovarian Tumors With the P53 Gene Mutation (MK-1775-004)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1775-004; 2011-002803-13 (EudraCT Number)
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Results first posted 2017-09-07 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — adavosertib; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1: adavosertib 225 mg + paclitaxel +carboplatin (Experimental): During the open-label run-in, participants receive 225 mg adavosertib twice daily (BID) starting on Day 1 of Cycle 1 (cycle=21 days) for a total of 5 doses. Participants receive adavosertib in combination with paclitaxel (175 mg/m2) and carboplatin (area under the curve [AUC] 5).
  Interventions: Drug: adavosertib; Drug: paclitaxel; Drug: carboplatin
- Part 2: adavosertib 225 mg + paclitaxel +carboplatin (Experimental): During Part 2, participants receive 225 mg adavosertib BID starting on Day 1 of each 21 day cycle for a total of 5 doses. Participants receive adavosertib in combination with paclitaxel (175 mg/m2) and carboplatin (AUC 5).
  Interventions: Drug: adavosertib; Drug: paclitaxel; Drug: carboplatin
- Part 2: Placebo + paclitaxel +carboplatin (Placebo Comparator): During Part 2, participants receive matched placebo to adavosertib BID starting on Day 1 of each 21 day cycle for a total of 5 doses. Participants receive placebo in combination with paclitaxel (175 mg/m2) and carboplatin (AUC 5).
  Interventions: Drug: Placebo; Drug: paclitaxel; Drug: carboplatin

INTERVENTIONS:
Drug: adavosertib — Adavosertib capsules, orally, twice a day (BID) for a total of 5 doses starting on Day 1 of each 3-week cycle
  Other Names: MK-1775
  Arms: Part 1: adavosertib 225 mg + paclitaxel +carboplatin; Part 2: adavosertib 225 mg + paclitaxel +carboplatin
Drug: Placebo — placebo to adavosertib, capsule, orally, BID for a total of 5 doses, starting on Day 1 of each 3-week cycle
  Arms: Part 2: Placebo + paclitaxel +carboplatin
Drug: paclitaxel — paclitaxel, intravenous (IV) infusion on Day 1 of each 3-week cycle
  Other Names: Taxol
Drug: carboplatin — carboplatin, IV infusion on Day 1 of each 3-week cycle
  Other Names: paraplatin

SUMMARY:
This is a study of the safety and efficacy of adavosertib in combination with paclitaxel plus carboplatin in the treatment of ovarian, fallopian tube, and primary peritoneal tumors with the P53 mutation. In Part 1, a small group of participants will receive adavosertib along with paclitaxel plus carboplatin to establish the tolerability of adavosertib with this combination. In Part 2, participants will be randomly assigned to receive either adavosertib plus paclitaxel and carboplatin OR placebo plus paclitaxel and carboplatin to assess efficacy of adavosertib compared to placebo. The primary hypothesis of the study (Part 2) is that administration of adavosertib in combination with paclitaxel plus carboplatin in participants with platinum sensitive p53 mutant ovarian cancer will result in improvement in progression free survival (PFS) per enhanced Response Evaluation Criteria In Solid Tumors version 1.1 (enhanced RECIST 1.1) compared to participants treated with paclitaxel plus carboplatin alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-low grade, non-borderline (low malignant potential) ovarian, fallopian tube, or primary peritoneal cancer which has progressed after paclitaxel / platinum-based therapy.
* Platinum-sensitive disease. Radiological progression must have occurred 6 months or more after the completion of the most recent platinum-based treatment.
* Measurable disease.
* Available tumor sample(s).
* Performance status of ≤1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Adequate organ function.

Exclusion Criteria:

* Pregnancy or the intention to become pregnant during the course of the study.
* Participation in a study with an investigational compound or device within 28 days of receiving first dose of study medication.
* Active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Primary CNS tumor.
* Known hypersensitivity or contraindications to the components of potential study therapy (paclitaxel, carboplatin, adavosertib) or its analogs (i.e., cremophor, mannitol, etc.).
* Participant requires the use of medications or products that are metabolized by, or inhibit, or induce Cytochrome P450 3A (CYP3A4).
* Ongoing peripheral neuropathies ≥Grade 2 and related to previous treatment.
* Known psychiatric or substance abuse disorders.
* Regular use (including "recreational use") of any illicit drugs or recent history (within the last year) of drug or alcohol abuse.
* HIV positive.
* Active Hepatitis B or C.
* Symptomatic ascites or pleural effusion.
* Clinical history suggestive of Li Fraumeni Syndrome.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2011-07-26 (Actual); Primary Completion 2016-08-08 (Actual); Study Completion 2016-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Fifteen participants were enrolled in Part 1 and 121 participants were enrolled in Part 2 (n=136 total).
Groups:
- Part 1: MK-1775 225 mg + Paclitaxel +Carboplatin: During the open-label run-in, participants received 225 mg MK-1775 twice daily (BID) starting on Day 1 of Cycle 1 (cycle=21 days) for a total of 5 doses. Participants received MK-1775 in combination with paclitaxel (175 mg/m^2) and carboplatin (area under the curve [AUC] 5).
- Part 2: MK-1775 225 mg + Paclitaxel +Carboplatin: During Part 2, participants received 225 mg MK-1775 BID starting on Day 1 of each 21 day cycle for a total of 5 doses. Participants received MK-1775 in combination with paclitaxel (175 mg/m^2) and carboplatin (AUC 5).
- Part 2: Placebo + Paclitaxel +Carboplatin: During Part 2, participants received matched placebo to MK-1775 BID starting on Day 1 of each 21 day cycle for a total of 5 doses. Participants received placebo in combination with paclitaxel (175 mg/m^2) and carboplatin (AUC 5).
Period: Part 1 (Open Label Run-in)
Arm/Group | Part 1: MK-1775 225 mg + Paclitaxel +Carboplatin | Part 2: MK-1775 225 mg + Paclitaxel +Carboplatin | Part 2: Placebo + Paclitaxel +Carboplatin
Started | 15 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 15 | 0 | 0
Not completed — Death | 5 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Study Terminated By Sponsor | 5 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Part 2 (Double-Blind Comparison)
Arm/Group | Part 1: MK-1775 225 mg + Paclitaxel +Carboplatin | Part 2: MK-1775 225 mg + Paclitaxel +Carboplatin | Part 2: Placebo + Paclitaxel +Carboplatin
Started | 0 | 59 (New participants enrolled in Part 2.) | 62 (New participants enrolled in Part 2.)
Treated | 0 | 59 | 60
Completed | 0 | 0 | 0
Not Completed | 0 | 59 | 62
Not completed — Death | 0 | 22 | 19
Not completed — Lost to Follow-up | 0 | 1 | 6
Not completed — Physician Decision | 0 | 1 | 4
Not completed — Progressive Disease | 0 | 1 | 3
Not completed — Study Terminated By Sponsor | 0 | 29 | 26
Not completed — Withdrawal by Subject | 0 | 5 | 4

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: MK-1775 225 mg + Paclitaxel +Carboplatin | Part 2: MK-1775 225 mg + Paclitaxel +Carboplatin | Part 2: Placebo + Paclitaxel +Carboplatin | Total
Number analyzed (Participants) | 15 | 59 | 62 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (9.9) | 58.3 (10.1) | 60.4 (9.8) | 59.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 59 | 62 | 136
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 2: Median Progression-free Survival (PFS) in Weeks Based on Enhanced Response Evaluation Criteria In Solid Tumors Version 1.1 (Enhanced RECIST 1.1) by Independent Radiology Review
Description: PFS was defined as the time from randomization to progressive disease (based on blinded independent central radiologic review) or death, whichever occurred earlier. Tumor response was evaluated every 6 weeks during treatment by diagnostic anatomic imaging and objective response assessments were performed based on enhanced RECIST 1.1 criteria. According to enhanced RECIST 1.1, progressive disease was the appearance of one or more new lesions, OR an unambiguous increase in the sum of target lesion volumes with both 1) >20% increase in the sum of volumes (SOV) of all target lesions (taking as reference the nadir) and 2) greater than two times the variability of the measurements estimated by the sponsor and/or its designees. PFS was analyzed for Part 2 participants only using the Kaplan-Meier method and median PFS was reported in weeks. Per protocol, Part 1 participants were not included in this analysis.
Time Frame: Up to 57 months
Population: Intent to Treat (ITT) Population: All randomized participants in Part 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part 1: MK-1775 225 mg + Paclitaxel +Carboplatin | Part 2: MK-1775 225 mg + Paclitaxel +Carboplatin | Part 2: Placebo + Paclitaxel +Carboplatin
Number analyzed (Participants) | 0 | 59 | 62
weeks |  | 34.14 [29.86 to 43.14] | 31.86 [24.43 to 35.57]
Statistical Analysis 1: Comparison: Part 2: MK-1775 225 mg + Paclitaxel +Carboplatin vs Part 2: Placebo + Paclitaxel +Carboplatin; A stratified [number of prior platinum based regimens (1 vs. 2 and 3), time since last platinum based therapy (<12 months vs. ≥12 months)] Cox proportional hazards model, with Efron method of tie handling, was used to assess the magnitude of the treatment difference between the treatment arms. The p-value from the score test was used in the significance test and the hazard ratio (MK-1775 versus Placebo) and its 95% confidence interval from the same Cox model was reported; Test type: Superiority or Other; p = 0.080, Cox proportional hazards model; Hazard Ratio (HR) = 0.63, 80% CI 2-sided [0.45 to 0.89]

2. Secondary Outcome: Part 1: Objective Response Rate (ORR) Per Gynecological Cancer Intergroup (GCIG) Criteria Based on Both RECIST 1.1 and Cancer Antigen 125 (CA-125) Level by Independent Radiology Review
Description: ORR was defined as the percentage of participants whose best response was confirmed partial response (PR) or complete response (CR) based both on imaging per RECIST 1.1 and on serum marker CA-125 level according to GCIC criteria. CR was defined by RECIST 1.1 as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have had reduction in short axis to <10 mm. PR was defined by RECIST 1.1 as at least a 30% decrease in the sum of the diameters (SOD) of target lesions, taking as reference the baseline SOD. A response according to CA-125 had occurred if there was ≥50% reduction in CA-125 levels from a pretreatment sample. The response must have been confirmed and maintained for at least 28 days. Participants could be evaluated according to CA-125 only if they had a pretreatment sample that was ≥2 times the upper limit of normal and within 2 weeks prior to starting treatment. Only evaluable Part 1 participants were included in this analysis.
Time Frame: Up to 57 months
Population: All participants receiving MK-1775 (225 mg) during Part 1 and evaluable at the time of the interim analysis. One participant took a prohibited medication during Part 1 and was considered unevaluable. Two participants enrolled into Part 1 after the interim analysis database lock and were not included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: MK-1775 225 mg + Paclitaxel +Carboplatin | Part 2: MK-1775 225 mg + Paclitaxel +Carboplatin | Part 2: Placebo + Paclitaxel +Carboplatin
Number analyzed (Participants) | 12 | 0 | 0
percentage of participants | 75.00 [42.814 to 94.514] |  |

3. Secondary Outcome: Part 2: Median PFS in Weeks Based on RECIST 1.1 by Independent Radiology Review
Description: PFS was defined as the time from randomization to progressive disease (based on blinded independent central radiologic review) or death, whichever occurred earlier. Tumor response was evaluated every 6 weeks during treatment by diagnostic anatomic imaging and objective response assessments were performed based on RECIST 1.1 criteria. According to RECIST 1.1, progressive disease was the appearance of one or more new lesions, OR a ≥20% increase in the sum of target lesion diameters (SOD) taking as reference the nadir (smallest SOD recorded since treatment started). PFS was analyzed for all randomized participants in Part 2 using the Kaplan-Meier method and median PFS was reported in weeks. Per protocol, Part 1 participants were not included in this analysis.
Time Frame: Up to 57 months
Population: ITT Population: All randomized participants in Part 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part 1: MK-1775 225 mg + Paclitaxel +Carboplatin | Part 2: MK-1775 225 mg + Paclitaxel +Carboplatin | Part 2: Placebo + Paclitaxel +Carboplatin
Number analyzed (Participants) | 0 | 59 | 62
weeks |  | 42.86 [35.00 to 48.86] | 34.86 [30.43 to 36.86]
Statistical Analysis 1: Comparison: Part 2: MK-1775 225 mg + Paclitaxel +Carboplatin vs Part 2: Placebo + Paclitaxel +Carboplatin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.030, Cox proportional hazards model; Hazard Ratio (HR) = 0.55, 80% CI 2-sided [0.39 to 0.79]

4. Primary Outcome: Part 1: Number of Participants With a Dose Limiting Toxicity (DLT)
Description: DLTs assessed during first 21-day cycle of Part 1 and defined as toxicities that met pre-defined severity criteria, were possibly, probably, or definitely related to triplet therapy, and could possibly result in a change in the given dose. Hematologic DLTs included Grade (Gr) 3 or Gr 4 neutropenia with fever >38.5°C and/or infection requiring antibiotic or anti-fungal treatment, and any Gr 4-5 hematological toxicity EXCEPT Gr 4 anemia, leukopenia, lymphopenia, neutropenia lasting <7 days, and thrombocytopenia lasting <4 days, except if a platelet transfusion was required. Non-hematologic DLT defined as any Gr 3, 4, or 5 nonhematologic toxicity EXCEPT: Gr 3 nausea, vomiting, diarrhea, or dehydration judged by Investigator and SPONSOR to occur in setting of inadequate compliance with supportive care measures and last for less than 48 hours, alopecia of any grade, inadequately treated hypersensitivity reactions, or clinically non-significant, treatable or reversible lab abnormalities.
Time Frame: During Cycle 1 of Part 1 (first 21 days)
Population: All participants who received ≥1 dose of study treatment during Cycle 1 of Part 1 open-label period and were evaluable at the time of the interim analysis. One participant took a prohibited medication during Part 1 and was considered unevaluable. Two participants enrolled into Part 1 after the interim analysis database lock and were not included.
Measure: Number; unit: participants
Arm/Group | Part 1: MK-1775 225 mg + Paclitaxel +Carboplatin | Part 2: MK-1775 225 mg + Paclitaxel +Carboplatin | Part 2: Placebo + Paclitaxel +Carboplatin
Number analyzed (Participants) | 12 | 0 | 0
participants
  Total | 3 |  |
  Febrile neutropenia | 1 |  |
  Neutropenia | 1 |  |
  Thrombocytopenia | 1 |  |

5. Primary Outcome: Parts 1 and 2: Percentage of Participants That Experienced an Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's products, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the SPONSOR's product was also an AE. The percentage of participants that experienced at least one AE was reported for each treatment arm.
Time Frame: Part 1: Day 1 through Post Study (286 days total). Part 2: Day 1 through Post Study (479 days total)
Population: Part 1: All participants who received at least one dose of study treatment during the open-label period.
  Part 2: All randomized participants who received at least one dose of study treatment. 2 participants were randomized to the Part 2 placebo arm but were not treated.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: MK-1775 225 mg + Paclitaxel +Carboplatin | Part 2: MK-1775 225 mg + Paclitaxel +Carboplatin | Part 2: Placebo + Paclitaxel +Carboplatin
Number analyzed (Participants) | 15 | 59 | 60
percentage of participants | 100.0 | 100.0 | 96.7
Statistical Analysis 1: Comparison: Part 2: MK-1775 225 mg + Paclitaxel +Carboplatin vs Part 2: Placebo + Paclitaxel +Carboplatin; P-values and 95% confidence intervals were calculated using the Miettinen and Nurminen method for between-treatment differences (MK-1775 vs. placebo) in the percentage of participants with events; Test type: Superiority or Other; Difference in Percentages = 3.3, 95% CI 2-sided [-2.9 to 11.4]

6. Primary Outcome: Parts 1 and 2: Percentage of Participants That Discontinued Study Treatment Due to an AE
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's products, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the SPONSOR's product was also an AE. The percentage of participants that discontinued study treatment (paclitaxel, carboplatin, or MK-1775) due to an AE was reported for each treatment arm.
Time Frame: Part 1: Day 1 through Post Study (286 days total). Part 2: Day 1 through Post Study (479 days total)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: MK-1775 225 mg + Paclitaxel +Carboplatin | Part 2: MK-1775 225 mg + Paclitaxel +Carboplatin | Part 2: Placebo + Paclitaxel +Carboplatin
Number analyzed (Participants) | 15 | 59 | 60
percentage of participants | 20.0 | 20.3 | 21.7
Statistical Analysis 1: Comparison: Part 2: MK-1775 225 mg + Paclitaxel +Carboplatin vs Part 2: Placebo + Paclitaxel +Carboplatin; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Difference in Percentages = -1.3, 95% CI 2-sided [-16.2 to 13.6]

7. Secondary Outcome: Part 2: ORR Per GCIG Criteria Based on Both Enhanced RECIST 1.1 and CA125 Level by Independent Radiology Review
Description: ORR defined as the percentage of participants with best response of confirmed PR or CR based both on imaging per enhanced RECIST 1.1 and on serum marker CA-125 level according to GCIC criteria. CR defined by enhanced RECIST 1.1 as disappearance of all target lesions. Any pathological lymph nodes (target or non-target) must have had reduction in short axis to <10 mm. PR was defined by enhanced RECIST 1.1 as ≥30% decrease in SOV of target lesions, taking as reference baseline SOV. Response according to CA-125 had occurred if there was ≥50% reduction in CA-125 levels from pretreatment sample. Response must have been confirmed and maintained for ≥28 days. Participants could be evaluated according to CA-125 only if they had a pretreatment sample that was ≥2 times the upper limit of normal and within 2 weeks prior to starting treatment. All randomized participants in Part 2 were analyzed. Per protocol, Part 1 participants were not included in this analysis.
Time Frame: Up to 57 months
Population: ITT Population: All randomized participants in Part 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: MK-1775 225 mg + Paclitaxel +Carboplatin | Part 2: MK-1775 225 mg + Paclitaxel +Carboplatin | Part 2: Placebo + Paclitaxel +Carboplatin
Number analyzed (Participants) | 0 | 59 | 62
percentage of participants |  | 74.58 [61.6 to 85.0] | 69.35 [56.3 to 80.4]
Statistical Analysis 1: Comparison: Part 2: MK-1775 225 mg + Paclitaxel +Carboplatin vs Part 2: Placebo + Paclitaxel +Carboplatin; Stratified Miettinen and Nurminen's method with a two-sided p-Value for testing was used for comparison of the ORRs between the treatment groups in Part 2 portion of the study. A 95% confidence interval (CI) for the difference in response rates was provided; Test type: Superiority or Other; p = 0.5247, Miettinen and Nurminen's Method; Difference in Response Rat = 5.2, 95% CI 2-sided [-10.9 to 21.1]

8. Secondary Outcome: Part 2: Median Overall Survival (OS) in Months
Description: OS was defined as the time from randomization to death due to any cause, reported in months. Participants without documented death at the time of analysis were censored at the date last known to be alive. For this endpoint, all randomized participants in Part 2 were analyzed. Per protocol, Part 1 participants were not evaluated for OS.
Time Frame: Up to 57 months
Population: ITT Population: All randomized participants in Part 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: MK-1775 225 mg + Paclitaxel +Carboplatin | Part 2: MK-1775 225 mg + Paclitaxel +Carboplatin | Part 2: Placebo + Paclitaxel +Carboplatin
Number analyzed (Participants) | 0 | 59 | 62
months |  | NA [20.34 to NA] — Median OS could not be calculated due to small percentage of death events observed by time of cut-off analysis date | NA [NA to NA] — Median OS could not be calculated due to small percentage of death events observed by time of cut-off analysis date
Statistical Analysis 1: Comparison: Part 2: MK-1775 225 mg + Paclitaxel +Carboplatin vs Part 2: Placebo + Paclitaxel +Carboplatin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.800, Cox proportional hazards model; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.40 to 3.34]

ADVERSE EVENTS:
Time Frame: Part 1: Day 1 through Post Study (286 days total). Part 2: Day 1 through Post Study (479 days total)
Description: Part 1: All participants who received at least one dose of study treatment during the open-label period (n=15).
  Part 2: All randomized participants who received at least one dose of study treatment (n=119). 2 participants were randomized to the Part 2 placebo arm but were not treated.
Arm/Group | Part 1: MK-1775 225 mg + Paclitaxel +Carboplatin | Part 2: MK-1775 225 mg + Paclitaxel +Carboplatin | Part 2: Placebo + Paclitaxel +Carboplatin
Serious Adverse Events (participants affected / at risk) | 9/15 | 24/59 | 12/60
Other Adverse Events (participants affected / at risk) | 15/15 | 59/59 | 57/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: MK-1775 225 mg + Paclitaxel +Carboplatin (N=15) | Part 2: MK-1775 225 mg + Paclitaxel +Carboplatin (N=59) | Part 2: Placebo + Paclitaxel +Carboplatin (N=60)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 13 (16) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 2 (4) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 2 (3) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 2 (2) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Medical observation (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: MK-1775 225 mg + Paclitaxel +Carboplatin (N=15) | Part 2: MK-1775 225 mg + Paclitaxel +Carboplatin (N=59) | Part 2: Placebo + Paclitaxel +Carboplatin (N=60)
Anaemia (Blood and lymphatic system disorders) | 6 (12) | 31 (68) | 19 (36)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 9 (25) | 12 (23)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 7 (16) | 24 (52) | 24 (58)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 21 (64) | 16 (31)
Palpitations (Cardiac disorders) | 1 (1) | 3 (4) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 3 (3) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1) | 5 (5) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 5 (5) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 2 (5) | 2 (2)
Diplopia (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 4 (4) | 2 (3)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 9 (11) | 14 (15)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 4 (9) | 2 (4)
Constipation (Gastrointestinal disorders) | 5 (5) | 17 (26) | 23 (29)
Diarrhoea (Gastrointestinal disorders) | 13 (34) | 44 (138) | 22 (39)
Dyspepsia (Gastrointestinal disorders) | 3 (5) | 6 (8) | 4 (5)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 3 (3) | 1 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 13 (27) | 46 (103) | 36 (67)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (2) | 1 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 8 (9) | 6 (7)
Vomiting (Gastrointestinal disorders) | 13 (33) | 37 (78) | 16 (19)
Asthenia (General disorders) | 2 (2) | 9 (16) | 2 (3)
Chills (General disorders) | 3 (5) | 3 (3) | 4 (7)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 13 (17) | 32 (54) | 33 (37)
Influenza like illness (General disorders) | 0 (0) | 3 (3) | 1 (1)
Injection site granuloma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 1 (1) | 1 (1)
Malaise (General disorders) | 3 (4) | 1 (1) | 4 (5)
Mucosal inflammation (General disorders) | 1 (1) | 3 (3) | 3 (3)
Oedema peripheral (General disorders) | 1 (3) | 9 (12) | 3 (3)
Peripheral swelling (General disorders) | 1 (1) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 7 (8) | 6 (7) | 6 (6)
Drug hypersensitivity (Immune system disorders) | 2 (4) | 6 (16) | 6 (8)
Hypersensitivity (Immune system disorders) | 1 (1) | 3 (4) | 4 (5)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 3 (3)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 4 (4)
Urinary tract infection (Infections and infestations) | 3 (6) | 7 (9) | 5 (7)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 6 (6) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 4 (4) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 2 (2) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (3) | 1 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 3 (6) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (8) | 12 (30) | 9 (34)
Platelet count decreased (Investigations) | 5 (9) | 8 (23) | 6 (20)
Weight decreased (Investigations) | 1 (1) | 2 (2) | 1 (1)
White blood cell count decreased (Investigations) | 5 (9) | 7 (17) | 6 (15)
Decreased appetite (Metabolism and nutrition disorders) | 8 (10) | 11 (18) | 11 (17)
Dehydration (Metabolism and nutrition disorders) | 5 (6) | 4 (10) | 3 (8)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 5 (15) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (5) | 8 (12) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (11) | 11 (16) | 9 (9)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (11) | 15 (20) | 16 (23)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 5 (5) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 15 (20) | 11 (17)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 6 (8) | 5 (8)
Dizziness (Nervous system disorders) | 4 (4) | 8 (15) | 7 (11)
Dysgeusia (Nervous system disorders) | 6 (9) | 9 (11) | 7 (15)
Headache (Nervous system disorders) | 2 (3) | 10 (11) | 8 (11)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 8 (9) | 9 (11)
Paraesthesia (Nervous system disorders) | 0 (0) | 3 (3) | 7 (9)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (9) | 12 (21) | 8 (9)
Polyneuropathy (Nervous system disorders) | 0 (0) | 6 (10) | 4 (5)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 3 (4) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 4 (5) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 3 (3) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (3) | 3 (4)
Depression (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (3) | 10 (13) | 8 (8)
Restlessness (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (3) | 2 (4) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 2 (2) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (2) | 0 (0) | 3 (3)
Urinary tract pain (Renal and urinary disorders) | 2 (3) | 1 (1) | 0 (0)
Breast oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (2) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 8 (10) | 6 (10)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 15 (23) | 8 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 4 (4) | 4 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (11) | 32 (33) | 40 (40)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (5) | 6 (6) | 7 (9)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2) | 5 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (8) | 4 (7) | 4 (4)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 3 (3) | 1 (1)
Flushing (Vascular disorders) | 4 (5) | 1 (3) | 4 (7)
Hypertension (Vascular disorders) | 5 (7) | 2 (2) | 3 (8)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication timelines.